CLINICAL TRIAL: NCT05008094
Title: The Epidemiology of Parkinson's Disease in Croatia and the Influence of Genetic Factors and Microbiota on the Progression and Treatment Outcomes of the Disease
Brief Title: The Epidemiology of Parkinson's Disease in Croatia and the Influence of Genetic Factors and Microbiota on the Progression and Treatment Outcomes of the Disease (GiOPARK)
Acronym: GiOPARK
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Clinical Hospital Center Rijeka (Other)
Collaborators: University Medical Centre Ljubljana (Other); Croatian Science Foundation (Other Government); Karolinska Institutet (Other)
Responsible Party: Sponsor
Other Study IDs: IP-2019-04-7276
Record Dates: First submitted 2021-08-04; First posted 2021-08-17 (Actual); Last update posted 2021-08-17 (Actual); Status verified 2021-08

CONDITIONS: Parkinson Disease; Genetic Disease; Microbiota; Neuro-Degenerative Disease; Neuroinflammatory Response
Keywords: Parkinson's disease; Genetics of Parkinson's disease; Microbiota; Microglia
MeSH Terms: conditions — Parkinson Disease; Genetic Diseases, Inborn | interventions — Exome; Magnetic Resonance Imaging; Electroencephalography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Genetic testing cohort (Phase 1): Group of Croatian Parkinson's disease patients who will be tested with whole-exome sequencing in target Parkinson's genes.
  Interventions: Diagnostic Test: Whole-exome sequencing
- Drug-naive Parkinson's disease patients (Phase 2): Drug-naive Parkinson's disease patients that will be prospectively followed in the two-year period for each patient.
  Interventions: Diagnostic Test: Whole-exome sequencing; Diagnostic Test: Microbiota sequencing; Diagnostic Test: Magnetic resonance imaging; Diagnostic Test: Transcranial ultrasound and Electroencephalography; Diagnostic Test: ELISA (Enzyme-Linked Immunosorbent Assay); Diagnostic Test: Fluorescent correlation spectroscopy (FCS)
- Control group (Phase 2): Control patients who do not have neurodegenerative diseases. The control group will perform the same measurement as the drug-naive Parkinson's disease patients.
  Interventions: Diagnostic Test: Whole-exome sequencing; Diagnostic Test: Microbiota sequencing; Diagnostic Test: Magnetic resonance imaging; Diagnostic Test: Transcranial ultrasound and Electroencephalography; Diagnostic Test: ELISA (Enzyme-Linked Immunosorbent Assay); Diagnostic Test: Fluorescent correlation spectroscopy (FCS)

INTERVENTIONS:
Diagnostic Test: Whole-exome sequencing — Whole-exome sequencing with the focus on Parkinson's disease loci.
Diagnostic Test: Microbiota sequencing — Next generation sequencing of microbiota from stool and saliva samples.
  Groups: Control group (Phase 2); Drug-naive Parkinson's disease patients (Phase 2)
Diagnostic Test: Magnetic resonance imaging — Magnetic resonance imaging of the brain focused on detection of free water in Substantia Nigra using a novel protocol.
  Groups: Control group (Phase 2); Drug-naive Parkinson's disease patients (Phase 2)
Diagnostic Test: Transcranial ultrasound and Electroencephalography — Transcranial ultrasound of Substantia Nigra, as well as high resolution EEG.
  Groups: Control group (Phase 2); Drug-naive Parkinson's disease patients (Phase 2)
Diagnostic Test: ELISA (Enzyme-Linked Immunosorbent Assay) — ELISA (Enzyme-Linked Immunosorbent Assay) will be used to assess the inflammatory state, glial functions, and disease progression will also be determined through specific markers in the participant's serum and plasma samples
  Groups: Control group (Phase 2); Drug-naive Parkinson's disease patients (Phase 2)
Diagnostic Test: Fluorescent correlation spectroscopy (FCS) — Fluorescent correlation spectroscopy (FCS), more specifically, ThT fluctuating intensity fluorescent analysis (FIFA) will be used to determine the existence of pathological conformation protein forms and their relation to the disease's grade and therapy.
  Groups: Control group (Phase 2); Drug-naive Parkinson's disease patients (Phase 2)

SUMMARY:
Parkinson's disease (PD) is the second most common neurodegenerative disease, which affects 2-3% of the general population above 65 years. There are significant differences in incidence depending on geographical location, race, and ethnicity. The exact cause of the disease is still unknown, but the role of genetic and environmental factors has already been established. Certain genetic forms of the disease make up for a small percentage, so it is thought that environmental factors have a more significant impact on the development of the disease. The incidence of PD is higher in people exposed to significant quantities of pesticides and traumatic brain injury, while there is a smaller incidence in smokers and people consuming more significant quantities of caffeine. The project will finish in four years, with the first 20 months dedicated to the first phase (genetic-epidemiological research), and the entirety of the 48 months for the second phase of the project (prospective clinical research).

The main goal of the first phase of the project is to determine which genetic mutations are the ones most represented in the Croatian population afflicted with the familial form of PD. In the second phase the main goal is to determine the influence of genetic factors and microbiological factors on the disease's progression as well as on the treatment outcomes. Specific goals of this part of the project are to determine how many patients in the general population of PD patients present with a genetic disorder and which genes have a role in that disorder, as well as determine the composition of intestinal and oral microbiota both in the patient test group and the healthy control group. Furthermore, specific goals are to evaluate the effects of standard PD treatment on the composition of microbiota, neurodegeneration progression and the activity of neuroinflammation in the central nervous system (CNS) and to examine whether there is a link between the physiological and the pathophysiological function of microbiota, using markers of disease progression and glial activity. Last specific goal is to analyze potential pathological conformation protein forms that could be used as a biomarker in early stages of the disease and a biomarker of disease progression.

The first phase of the study will provide the first epidemiologic data on the familial form of PD, as well as the mutations most represented in patients with PD in Croatia. Additionally, the prospective clinical study will contribute to enlightening the intertwined effects of genetic and environmental factors in the emergence and progression of the disease, as well as their effect on treatment outcome. Intestinal and oral microbiota composition analysis will determine whether there is a difference between PD and the healthy population while using the short-chain fatty acid profile will determine the metabolic differences between the two groups. Analyzing the markers of CNS homeostasis, inflammation, and neuroglial function will determine the progression of the disease and also correlate them to genetic factors as well as the microbiota function and composition. Analyzing the pathological conformation forms of alpha-synuclein could lead to the discovery of novel biomarkers in the early stages of the disease, as well as to follow the progression of the disease

DETAILED DESCRIPTION:
Parkinson's disease (PD) is the second most common neurodegenerative disease, which affects 2-3% of the general population above 65 years. There are significant differences in incidence depending on geographical location, race, and ethnicity. The exact cause of the disease is still unknown, but the role of genetic and environmental factors has already been established. Certain genetic forms of the disease make up for a small percentage, so it is thought that environmental factors have a more significant impact on the development of the disease. The incidence of PD is higher in people exposed to significant quantities of pesticides and traumatic brain injury, while there is a smaller incidence in smokers and people consuming more significant quantities of caffeine.

Moreover, intestinal and oral microbiota is regarded as a significant factor in the pathogenesis of the disease, due to the discovered floral imbalance in people suffering from PD. At this point, it is unknown whether the dysbiosis of the intestinal microbiota precedes the disease or it is the result of the disturbed neuronal communication of the liver-brain axis. Since there has not been a proper epidemiological study conducted in Croatia so far, there is no knowledge of the number of cases of PD linked with genetic and environmental factors, doing this project that more scientifically and socially impactful.

A specific pathophysiological event in PD is the loss of neurons in the substantia nigra, along with the accumulation of the intracellular protein α-synuclein in the entire central nervous system. It is important to note that PD is asymptomatic for an extended period since the symptoms start manifesting only when there is a loss of more than 70-80% of dopaminergic neurons. Dysfunction of glial cells, cells that are usually in charge of keeping homeostatic conditions in the central nervous system accompanies PD. The dysfunction leads to neuroinflammation and microglial activation, phagocytosis and the destruction of neurons. On the other hand, there is a lack of a proper nutritive and reparative reaction from astrocytes, glial cells involved in neuroprotection and injury repair in the CNS. Unfortunately, there is still no specific biomarker known for PD, however alterations of neurodegenerative, nutritive, and immunological markers in these disorders enable experimental monitoring of disease progression. Recent research proposed a link between intestinal microflora and glial cells in physiological conditions, but also in the pathogenesis of various neurodegenerative disorders. It is currently thought that the first pathophysiological changes, occur inside the intestinal nervous system, which is in direct contact with the intestinal microflora. This way the intestinal microbiota could modulate the pathogenesis of PD and contribute to the interindividual variability of the clinical presentation. Even though a small number of studies did focus on this part of the pathogenesis of the disease, the real effect of the intestinal and oral microflora dysbiosis on the pathogenesis of PD is not established. Also, there have been no studies which explore the relationship between genetic and environmental factors, making prospective studies with de novo PD patients necessary in shedding light on the mean effects of the dysbiosis on the disease progression and treatment outcome.

The project will finish in four years, with the first 20 months dedicated to the first phase (genetic-epidemiological research), and the entirety of the 48 months for the second phase of the project (prospective clinical research) Participants: The research group in the first phase of the research includes patients with PD throughout the Republic of Croatia. The population would include all the available afflicted currently residing in Croatia, which are members or work with the Croatian PD patient's association. The estimated response is 10% of the PD population (500-750 patients) The patients will fill the epidemiologic questionnaires and patients with familial PD will be selected. The expected emergence of the hereditary form of the disease in the PD population is around 10-15% (50-75). The second phase of the research (prospective clinical trial) includes two subject groups. The first will be made up from patients from the Clinical Hospital Centers in Rijeka, which have not been actively treated yet (drug-naive), while the second will consist of healthy controls in the same age range. The target number of subjects in both of these two groups is 50. Inclusion criteria for participation of drug-naïve patients is a confirmed PD diagnosis according to the Movement Disorder Society Clinical Diagnostic criteria. The healthy control group will consist of participants from the same age group with the same nutritional status (body mass index), as well as living in the same geographical area as the test group. Exclusion criteria for participation include unique diet plans, chronic bowel disease, any autoimmune disorder, acute infectious diseases, acute active inflammation, patient history positive for significant gastrointestinal surgical procedures and an active antibiotic, probiotic, nutritive supplement, corticosteroid, and immunosuppressive drugs.

The first phase - genetic-epidemiological study (20 months): In the first nine months, throughout Croatia, participants who are members or work with the Croatian PD patient's association will be recruited. At the end of the first year of the research, the participants will have their whole exomes sequenced with the help of next-generation sequencing (NGS), to find genetic variants in Croatian patients. Through the second year of research, result analysis and dissemination are planned, as well as counseling in participants with a confirmed familial variant of the disease. For this purpose, the participants will give blood samples for genetic analysis. The target number of subjects in this phase of the research is 50. The participants will also be asked to fill out several structured study forms, which should provide an estimation of the genetic background of the participant, along with information on their biorhythm, sleep patterns, diet, life goals, and general stress.

The second phase - a prospective clinical study (48 months): Participant selection will be conducted throughout the first year of the clinical study. The following time intervals are selected for control visits: baseline; 6 months, 12 months, 24 months and 30 months. The result analysis and dissemination are planned in the last two years of research. Every participant in the study will have their exome sequenced with NGS, with the focus mostly being on parts that have a known impact on the pathogenesis of PD. Both the patients and healthy control population will also have their microbiota composition determined with NGS, as well as their functional state through the analysis of the short-chain fatty acid composition, known metabolic products of the microbiota. ELISA (Enzyme-Linked Immunosorbent Assay) will be used to assess the inflammatory state, glial functions, and disease progression will also be determined through specific markers in the participant's serum and plasma samples. Fluorescent correlation spectroscopy (FCS), more specifically, Thioflavin T (ThT) fluctuating intensity fluorescent analysis (FIFA) will be used to determine the existence of pathological conformation protein forms and their relation to the disease's grade and therapy. It is for these methods that the participants will be asked to give a blood, stool, and saliva sample. The disease progression will also be monitored with transcranial B-mod sonography and magnetic brain resonance.

The exome sequencing will be conducted at baseline, while the analysis of the composition and function of microbiota will be performed on the first and last control visit. Biomarker analysis, protein conformation analysis and neuro-radiological methods will be conducted at every control examination. From the first visit, the participants will be asked to fill out several structured study questionnaires, which will provide an estimation of the genetic background of the participant, along with information on their biorhythm, sleep patterns, diet, life goals, and general stress. Moreover, the cognitive state of the participants will be evaluated through validated tests like the Mini-Mental State Examination (MMSE) and the Montreal Cognitive Assessment (MoCA), while the general non-motoric symptoms will be evaluated with the help of the Non-Motor Symptoms Questionnaire (NMSQ) and the Non-Motor Symptoms Scale (NMSS). Patients will also be evaluated with the help of the UPDRS (Unified Parkinson's disease rating scale), the most prominently scale in PD.

The main goal of the first phase of the project is to determine which genetic mutations are the ones most represented in the Croatian population afflicted with the familial form of PD. In the second phase the main goal is to determine the influence of genetic factors and microbiological factors on the disease's progression as well as on the treatment outcomes. Specific goals of this part of the project are to determine how many patients in the general population of PD patients present with a genetic disorder and which genes have a role in that disorder, as well as determine the composition of intestinal and oral microbiota both in the patient test group and the healthy control group. Furthermore, specific goals are to evaluate the effects of standard PD treatment on the composition of microbiota, neurodegeneration progression and the activity of neuroinflammation in the CNS and to examine whether there is a link between the physiological and the pathophysiological function of microbiota, using markers of disease progression and glial activity. Last specific goal is to analyze potential pathological conformation protein forms that could be used as a biomarker in early stages of the disease and a biomarker of disease progression.

The first phase of the study will provide the first epidemiologic data on the familial form of PD, as well as the mutations most represented in patients with PD in Croatia. Additionally, the prospective clinical study will contribute to enlightening the intertwined effects of genetic and environmental factors in the emergence and progression of the disease, as well as their effect on treatment outcome. Intestinal and oral microbiota composition analysis will determine whether there is a difference between PD and the healthy population while using the short-chain fatty acid profile will determine the metabolic differences between the two groups. Analyzing the markers of CNS homeostasis, inflammation, and neuroglial function will determine the progression of the disease and also correlate them to genetic factors as well as the microbiota function and composition. Analyzing the pathological conformation forms of alpha-synuclein could lead to the discovery of novel biomarkers in the early stages of the disease, as well as to follow the progression of the disease

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria for participation of drug-naïve patients is a confirmed PD diagnosis according to the Movement Disorder Society Clinical Diagnostic criteria.
* The healthy control group will consist of participants from the same age group with the same nutritional status (body mass index), as well as living in the same geographical area as the test group.

Exclusion Criteria:

* unique diet plans, chronic bowel disease, any autoimmune disorder, acute infectious diseases, acute active inflammation, patient history positive for significant gastrointestinal surgical procedures and an active antibiotic, probiotic use.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The research group in the first phase of the research includes patients with PD throughout the Republic of Croatia. The population would include all the available afflicted currently residing in Croatia, which are members or work with the Croatian PD patient's association. The estimated response is 10% of the PD population (500 patients). The patients will fill the epidemiologic questionnaires and patients with confirmed PD in the family will be selected. The expected emergence of the hereditary form of the disease in the PD population is around 10-15% (500-750).
  The second phase of the research (prospective clinical trial) includes two subject groups. The first will be made up from patients from the Clinical Hospital Centers in Rijeka and Zagreb, which have not been actively treated yet (drug-naive), while the second will consist of healthy controls in the same age range. The target number of subjects in both of these two groups is 50.
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2020-05-01 (Actual); Primary Completion 2023-08-01 (Estimated); Study Completion 2024-02-01 (Estimated)

PRIMARY OUTCOMES:
Genetic mutations in familial or early onset Croatian Parkinson's disease patients | 20 months
  Determining which genetic mutations are the ones most represented in the Croatian population afflicted with the familiar or early onset form of PD.
Influence of genetic factors on the disease's progression and treatment outcomes. | 48 months
  Determining the influence of genetic factors on the disease's progression and treatment outcomes.
Influence of microbiological factors on the disease's progression and treatment outcomes. | 48 months
  Determining the influence of microbiological factors on the disease's progression and treatment outcomes.

SECONDARY OUTCOMES:
Genetic factors in general Croatian Parkinson's disease patients | 48 months
  determining how many patients in the general population of PD patients are linked with genes and which genes have a role in that disorder.
Composition of microbiota in Croatian PD patients and controls | 48 months
  Determining the composition of intestinal and oral microbiota both in the patient test group and the healthy control group.
Effects of Parkinson's disease treatment on microbiota and inflammatory response in Parkinson's disease patients | 48 months
  Evaluating the effects of standard PD treatment on the composition of microbiota, neurodegeneration progression and the activity of neuroinflammation in the CNS.
Influence of microbiota and inflammatory factors on progression and treatment in Croatian PD patients | 48 months
  Examining whether there is a link between the physiological and the pathophysiological function of microbiota, using markers of disease progression and glial activity.
Pathological alpha-synuclein conformation in PD patients and controls | 48 months.
  Analyze potential pathological conformation protein forms that could be used as a biomarker in the early stages of the disease and a biomarker of disease progression

CONTACTS AND LOCATIONS:
Overall Officials: Vladimira Vuletic, Principal Investigator — Clinical Hospital Center Rijeka
Locations (1):
- Clinical Hospital Center Rijeka, Rijeka, Croatia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Project website — https://neurolab.uniri.hr/?page_id=2